CLINICAL TRIAL: NCT06315192
Title: Stroke Alarm Efficacy Trial
Acronym: StrokeAlarmEFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Karolinska University Hospital (Other); Stockholm South General Hospital (Other); Sahlgrenska University Hospital (Other); Skane University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CIV-22-10-041006
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Stroke Acute; Atrial Fibrillation; TIA
Keywords: Stroke; wearable; indication; sensor
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective observational single-arm trial with a registry-based propensity matched control population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke Alarm use (Experimental): The patients are provided with Stroke Alarm and instructed to use it in accordance with the IFU for a 3 months period.
  Interventions: Device: Stroke Alarm

INTERVENTIONS:
Device: Stroke Alarm — Patients who meet the criteria for participation will, after signing consent, be included and receive the Stroke Alarm bracelets that are used for 3 months. Study data will be collected as baseline at inclusion, at follow-up 3 months after inclusion and by using national Swedish registry data after completion of the study.

SUMMARY:
The aim of this study is to test the efficacy of the CE-marked wearable system Stroke Alarm to identify the onset of a stroke with unilateral arm motor deficit within 3 hours of onset.

This is a multicenter, prospective observational single-arm trial with a registry-based propensity matched control population.

A total of 500 patients will be included in the trial. An interim analysis will determine if the stroke onset frequency is sufficient to determine the main outcome. Should the number of stroke events differ from what is expected at interim analysis, study enrollment will continue to increase cohort size.

Patients who meet the criteria for participation will, after signing consent, be included and receive the Stroke Alarm bracelets that are used for 3 months. Study data will be collected as baseline at inclusion, at follow-up 3 months after inclusion and by using national Swedish registry data after completion of the study.

Patients with elevated stroke risk according assessed by presence of specific criteria associated with elevated risk caused by:

1. recent TIA, OR
2. recent stroke without persisting arm motor deficit, OR
3. atrial fibrillation A control population matched for age, sex, NIHSS score and health care region will be identified in the Swedish national stroke registry, Riksstroke, and used for comparison.

The combined efficacy goal is at least 60% sensitivity for Stroke Alarm b of stroke with unilateral arm motor deficit within 3 hours of onset (with a 95% confidence interval above 30%) and a specificity of at least 80% using a clinical stroke diagnosis as gold standard.

DETAILED DESCRIPTION:
Objectives and hypotheses of the clinical investigation The aim of this study is to test the ability and efficacy of the CE-marked wearable system Stroke Alarm to detect a stroke onset early.

The hypothesis is that the Stroke Alarm is able to indicate at least 60% of stroke cases with unilateral arm motor deficit within 3 hours of onset with a specificity of at least 80%.

Design of the clinical investigation This is a prospective single arm observational trial with a propensity-matched registry-derived control group.

All patients with a diagnosis of stroke (ischemic stroke or intracerebral hemorrhage) without arm motor deficits, TIA or atrial fibrillation at the participating hospitals that fullfill all inclusion critera and no exclusion criteria is asked for participation in the trial.

The patient is after the setup wearing the device continuously for three months.

An administrative follow-up is performed at 90-120 days following inclusion, the EPR is reviewed for any hospital admissions for stroke during the study period.

No standard care comparator will be used in this study, mainly because of lack of similar systems to compare with and blinding issues.

Simultaneous inclusion in other studies that require bracelets are not permitted, but inclusion in other clinical treatment trials, such as for drugs och medical devices that does not require bracelets, are acceptable.

Study population All patients (age ≥ 60 years) with a diagnosis of stroke (ischemic stroke or intracerebral hemorrhage) without arm motor deficits, TIA or atrial fibrillation at the participating hospitals is candidates for participation in the trial.

Enrollment Patients with a diagnosis of stroke (ischemic stroke or intracerebral hemorrhage) without arm motor deficits, TIA or atrial fibrillation that fullfill all inclusion and no exclusion criteria are included after signing the informed consent form at inclusion visit after oral and written information within the hospital or at an out-patient facility (described in Informed consent process, section 16).

Included subjects are added to the identification log stored in the Investigators Site File (ISF) that is located in locked research offices at the participating hospitals. The Identification log is under no circumstances shared or moved from the ISF that is located at participating hospital.

The patients are instructed to use the device continuously for three months. When setting-up the app on their smartphones they will be required to add at least one alarm recipient, but adding more alarm recipients is encouraged. The recipients are independent of study design and can be family members, friends or neighbors, as preferred by the subjects.

Device startup The study nurses manage the inclusion procedure that are recorded in the EPR and the administrative system according to the local regulations of the including center.

The wearable stroke indication system is given to the patient when accepting inclusion in the trial. The system will include a user manual with step-by-step instructions that are used during the activation of the investigational device, Stroke Alarm. The Study nurse may also assist in activation, including adding alarm recipients which is exactly the same as expected during clinical routine use.

The product is designed for continuous use for up to 6 months in a home environment and can also be used in a hospital environment. The devices will not be re-used for another subject and collected by the manufacturer at the end of the study.

The device is not MR-compatible. The included patient is the user of the device. Each participant will receive one unit of Stroke Alarm, consisting of a pair of sensor bracelets and one IFU. The smartphone app is downloaded from Apple's AppStore (iOS) or via Google Play (Android). Other operative systems can't be used.

The device is intended to be used continuously during the entire study period of 90 days. During the study the user is instructed to use the device according to the IFU. The user is instructed to use the device in his/her regular activities in the home environment continuously during the entire study period.

For the device to be fully functional, the user needs to activate and wear both sensor bracelets, install the Stroke Alarm app, complete the on-boarding and have at least one alarm recipient who has accepted the invitation to act as alarm recipient. Also, for the device to be fully functional, the user needs to be within Bluetooth connection from his/her smartphone, the smartphone needs to be active and have wifi- or 3G/4G/5G internet access.

At startup, the user invites Alarm recipients, who will be alerted via SMS messages in case the device indicates stroke by identifying arm motor deficiency that may be consistent with stroke and the initial indication is not abolished by the user. Any number of Alarm recipients can be chosen, typically they may be relatives, neighbors and friends. An Alarm recipient is not registered to the system unless he/she accepts his/her role as an Alarm recipient for the user. At least one confirmed Alarm recipient is necessary for the system to be operational. Alarm recipients can be added or removed during the study period. The choice of, and role for the Alarm recipients is identical in the study as in regular use. That means that the user will select Alarm recipients based on his/her own preferences and they are supposed to react to any alarms from the device as they would to the device in regular use. An Alarm recipient is not a study subject, and no informed consent is obtained. The identity of the Alarm recipients is not collected in the study.

During setup are the user testing the stroke test (Appendix A) that consists of 8 questions/tasks designed to mimic the items tested by the NIHSS and the different types of sound and/or vibration alarms (described below and appendix??) for better understanding of the differences between them.

Similar to regular use of the device, the study subjects may contact the manufacturer's support-service for questions and support related to the device.

Alarm description A false indication is an indication made by the algorithm from imbalance of arm activity in the absence of a stroke. It can occur during everyday activity dominated by one arm. It will lead to a false alarm if it is not abolished by user tests.

Dedicated arm motion (Escalation step 1, Figure 2) is a specified gesture ("draw a ball in the air") that is used to identify erroneous indications.

In-app test (Escalation step 2, Figure 2) is the test included in the Stroke Alarm smartphone app intended to abolish erroneous indications that are not eliminated by a dedicated arm motion (Escalation step 1).

A false alarm is a SMS alarm sent to the Alarm recipients based on an initial false indication made by the algorithm in the absence of a stroke with unilateral arm motor defecit.

SMS messages to the Alarm recipients generated by technical problems that affect the function of the device (for example loss of internet-connection or loss of Bluetooth-connection) is not considered false alarms.

If the user suffers a stroke and is not able to alert himself/herself and an arm paresis associated with the stroke is detected by the device, this will first generate a true indication manifested as vibration in the bracelet of the affected arm. If the user does not abolish this indication by a dedication arm movement, it will trigger a local alarm in the smartphone within 30 seconds. If the user does not open the smartphone app and complete the in-app stroke test within 10 minutes a SMS alarm is sent to all Alarm recipients. Alarm recipients are then expected to promptly act to ensure that the user is either confirmed to be well or is taken care of by healthcare, similar as if the user had called for help by any other means.

If the user suffers a stroke with unilateral arm weakness and is not able to alert himself/herself and no arm paresis is detected by the device (false negative) the device have not contributed to patient care and stroke diagnosis, similar to if the device not was present. In this case the workflow is the same as without the device; which means that the patient will need to alert healthcare himself/herself, of by help of others who may be present at onset or who may discover the patient at a later timepoint.

The device does not contact health care services. This contact must be initiated by the user or by Alarm recipients alerted by the device or other means.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 50 years or older
2. Modified Rankin scale of 0-2.
3. Diagnosed with either:

   A. Recent* transient ischemic attack (TIA, G45.9), AND:
   * ABCD2 score of ≥6, OR:
   * Atrial fibrillation OR:
   * Large artery atherosclerosis**.

   B. Recent* acute ischemic stroke (I63), AND:

   • Atrial fibrillation, OR:
   * Large artery atherosclerosis**. C. Atrial fibrillation/flutter (I48), AND
   * None, or reduced dose of, oral anticoagulation medication***, AND
   * CHA2DS2-VASC score ≥4.

   D. Recent* intracerebral hemorrhage (I61.9), AND:

   • Atrial fibrillation.
4. The patient has received the required information about the study and agrees in writing to participate.
5. Smartphone user since at least 1 year.

   * Within the last 2 weeks **Atherosclerosis in carotid, vertebral aortic arch or major intracerebral arteries according to CTA or ultrasound.

     * Including all oral anticoagulation medication such as Warfarin and NOACs. Patients with reduced dose of a NOAC can be included, regardless if this is within the approved label, or if reduced dose is chosen off-label for other reasons. Treatment with antiplatelet medication is permissible.

EXCLUSION CRITERIA

1. Previous inclusion in this study.
2. Arm motor deficit from any previous medical condition.
3. Unable to give informed consent to participate in the study.
4. Does not master any of the languages available within the Stroke Alarm smartphone app in speech and writing.
5. Does not have access to a Stroke Alarm compatible smartphone.
6. Deemed unable to handle the Stroke Alarm smartphone app, or participate in planned follow-up within the framework of the study due to other diseases or circumstances.
7. Does not want to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time from onset of stroke with unilateral arm motor deficit until alarm by the device. | An alarm generated within 3 hours following onset of stroke with unilateral arm paresis
  The alarm is recorded systematically from the device backend. The ground truth is gathered based on the medical records for stroke events during the study period. Pre-set definitions are defined what is considered a true positive, a false positive, a true negative and a false negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Anderson, Ms., Study Director — Lund University
Locations (5):
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Hässleholms sjukhus, Hässleholm
  - Karolinska University Hospital Huddinge, Huddinge
  - Skane University hospital, Lund
  - Skåne University Hospital Malmö, Malmo

IPD SHARING:
Plan to Share IPD: Undecided